CLINICAL TRIAL: NCT02209246
Title: The Effect of Feedback Regarding Illness Behavior on Patient Satisfaction in Hand Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David C. Ring, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Purpose: Health Services Research
Other Study IDs: 2013P001425
Record Dates: First submitted 2014-07-29; First posted 2014-08-05 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Hand Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The intervention group will be comprised of patients who will complete the PROMIS- CAT for pain interference, pain behavior and physical function prior to the encounter with the physician and then will complete the MISS-21 after the encounter.
  Interventions: Other: PROMIS CAT Pain Interference; Other: PROMIS CAT Pain Behavior; Other: PROMIS CAT Physical Function; Other: MISS-21
- Control (Experimental): The control group will complete the PROMIS- CAT for pain interference, pain behavior and physical function after the encounter and after completing a satisfaction questionnaire (MISS-21).
  Interventions: Other: PROMIS CAT Pain Interference; Other: PROMIS CAT Pain Behavior; Other: PROMIS CAT Physical Function; Other: MISS-21

INTERVENTIONS:
Other: PROMIS CAT Pain Interference
Other: PROMIS CAT Pain Behavior
Other: PROMIS CAT Physical Function
Other: MISS-21

SUMMARY:
The investigators of this study would like to see whether providing feedback to patients regarding their illness behavior/coping strategies, using online questionnaires, improves patient-physician communication in orthopaedic surgery. The investigators aim to enroll 128 patients.

DETAILED DESCRIPTION:
Psychological and sociological factors are important in the human illness experience, but biomedical factors are the focus of most office visits, particularly in hand surgery. Both patients and surgeons can feel uncomfortable discussing emotions, stress, and coping strategies. Detmar et al. randomized patients in an oncology practice to receive feedback on a HRQL assessment or not during office visits. They observed that feedback on the HRQL assessment contributed to physicians' awareness of healthy issues and patient-physician communication. There was a difference in perceived emotional support, but not in overall satisfaction with the visit[1]. A retrospective study observed in patients with local prostate cancer, that pre-therapy HRQL assessment is associated with a better sexual function, sexual bother and bowel function according to post-therapy HRQL scores[2].

The investigators propose a two arm unblended, randomized (1:1) controlled trial to assess the effect of providing feedback to patients regarding illness behavior/coping strategies (using Patient Reported Outcomes Measurement Information System (PROMIS) Computer Adaptive Testing (CAT) instruments) on patient satisfaction and patient-physician communication in orthopaedic surgery.

If the results of the study suggest that feedback of results from the questionnaires increases patients' satisfaction, such an intervention may be used in the future to benefit future patients.

Aim:

The aim of this study is to assess the effect of feedback regarding illness behavior measured with Patient Reported Outcomes Measurement Instrument System - Computerized Adaptive Testing (PROMIS- CAT) on patient satisfaction.

Primary Null Hypothesis:

There is no difference in satisfaction between patients who receive feedback about their illness behavior, measured with PROMIS-CAT, compared to patients who do not.

Secondary Null Hypotheses:

There is no difference in patient-physician communication about patient's illness behavior between patients who receive feedback about their illness behavior, measured with PROMISCAT, compared to patients who do not.

There are no predictors for patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* All new patients visiting the Orthopaedic Hand and Upper Extremity Service
* English fluency and literacy
* Ability to provide informed consent

Exclusion Criteria:

* age < 18
* Inability to complete enrollment forms due to any mental status or language problems (e.g. dementia, head injury, overall illness).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2013-07; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
PROMIS CAT Pain Interference | 1 day
  A computerized assessment of pain interference measured at enrollment
PROMIS CAT Pain Behavior | 1 day
  A computerized assessment of pain behavior measured at enrollment
PROMIS CAT Physical Function | 1 day
  A computerized assessment of physical function measured at enrollment
Medical Interview Satisfaction Scale (MISS-21) | 1 day
  Questionnaire

SECONDARY OUTCOMES:
Patient-physician communication | 1 day
  The research assistant determines whether the patient's coping strategies (pain interference and pain behavior) were discussed during the encounter or not.

CONTACTS AND LOCATIONS:
Overall Officials: David Ring, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Detmar SB, Muller MJ, Schornagel JH, Wever LD, Aaronson NK. Health-related quality-of-life assessments and patient-physician communication: a randomized controlled trial. JAMA. 2002 Dec 18;288(23):3027-34. doi: 10.1001/jama.288.23.3027. PMID 12479768
- [Background] Chamie K, Sadetsky N, Litwin MS. Physician assessment of pretreatment functional status: a process-outcomes link. J Urol. 2011 Apr;185(4):1229-33. doi: 10.1016/j.juro.2010.11.087. Epub 2011 Feb 22. PMID 21334026